CLINICAL TRIAL: NCT06612996
Title: Comparative Study Between Intravenous Tramadol and Magnesium Sulphate for Prevention of Shivering Post Intrathecal Anesthesia a Randomized Clinical Study
Brief Title: Intravenous Tramadol and Magnesium Sulphate for Prevention of Shivering
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Warda Demerdash Khalifa Ali, Dr, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AZAST/19/14-May-2024
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Lower Extremity Chronic Venous Ulcers; Varicose Veins Leg; Hernia
Keywords: Tramadol; Magnesium Sulphate; Shivering
MeSH Terms: conditions — Hernia | interventions — Tramadol; Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tramadol group (Experimental): Intravenous Tramadol
  Interventions: Drug: Tramadol
- Magnesium sulphate group (Experimental): Intravenous Magnesium Sulphate
  Interventions: Drug: Magnesium sulphate
- Control group (Placebo Comparator): Saline
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Tramadol — Intravenous tramadol
  Arms: Tramadol group
Drug: Magnesium sulphate — Intravenous magnesium sulphate
  Arms: Magnesium sulphate group
Other: Saline — Normal saline
  Arms: Control group

SUMMARY:
The aim of this work was to compare the efficacy of intravenous (IV) tramadol versus magnesium sulphate added to 100 ml saline for prevention of shivering associated with spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

- American Society of Anesthesiologists (ASA) I and II physical status undergoing an elective surgery under spinal anesthesia.

Exclusion Criteria:

* history of uncontrolled comorbidities, cardiac, respiratory, renal or hepatic disease, patients who had allergy to any medication in the study, contraindications to spinal anesthesia (coagulation disorder, infection at site of puncture, raised intracranial tension or any spine deformity), fever >38 Celsius or less than 36 Celsius, body mass index more than 35 and who has history of alcohol intake

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Shivering score | 90 minutes postoperatively
  Shivering score

IPD SHARING:
Plan to Share IPD: No